CLINICAL TRIAL: NCT02467205
Title: Effectiveness of Community Based Physical Activity on Step Count and Sedentary Behaviour in Patients With Rheumatoid Arthritis Within the First Five Years of Diagnosis
Brief Title: Walk for Rheumatoid Arthritis (WARA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Amal Elramli, PhD student and chief investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GN14RH210
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Physical Activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): pedometer supported walking and education A ;pedometer will be given to each person in the intervention group at the first education session. Participants will be encouraged to use the pedometer for a 6 month period Educational component; participants will attend six weekly sessions in small groups of up to six people; the content of the sessions will be based on educational cognitive behavioural programme development, In addition, participants will receive education material in the first education session. The intervention group will receive two booster sessions, after 3 and 6 months.
  Interventions: Other: pedometer supported walking and education
- Control (No Intervention): participants randomly allocated to the comparison group will receive one education session (visit 2) regarding the importance of exercise and healthy diet and will be given education material similar to intervention group and encouraged to read it.

INTERVENTIONS:
Other: pedometer supported walking and education — A Physical activity; pedometer will be given to each person in the intervention group at the first education session. Participants will be encouraged to use the pedometer for a 6 month period.
  The strength exercises will be performed at home. Education will incorporate the behavioural change techniques (BCTs) known to be effective in increasing physical activity (Goal setting,Self-monitoring of behaviour,Feedback on outcomes of behaviour,Problem solving,Relapse Prevention (RP) and social support).
  Arms: Intervention

SUMMARY:
The overall aim of this randomized control trial study is to investigate the effectiveness of a six-month, community based, pedometer supported, walking programme, along with an education programme incorporating behavioural change techniques on steps count and sedentary time, disease activity, functional capacity and cardiovascular risk of people within the first five years of being diagnosed with RA.

DETAILED DESCRIPTION:
All patients attending the rheumatology clinics at Gartnavel General Hospital, Glasgow Royal Infirmary and Stobhill Hospital who have received a diagnosis of rheumatoid arthritis, according to the American College of Rheumatology revised Criteria (ACR) 1987/European League Against Rheumatism (EULAR) 2010 (Amett et al, 1988; Aletaha et al, 2010) within the first five years of disease will be eligible to take part. Patients will be informed of the study at their routine clinical appointments and will be given study information sheets, in order to inform and help them decide whether they would like to enroll in the study. If the patient is willing to take part in the study, they will contact the researcher by phone and a suitable date/time for assessment will be arranged and confirmed by letter. For further enquiries, patients can telephone the researcher via contact details on the study information sheet. All participants will be informed that they are free to withdraw from the study at any time. On the initial assessment day, the participant will have the opportunity to ask further questions before being asked to sign a consent form for the study. All participants who agree to take part will be required to consent to being randomized to either the physical activity (Walking) group; Group (1) or Comparison group; Group (2).

A pedometer will be given to each person in the intervention group at the first education session.Participants will be encouraged to use the pedometer for a 6 month period, and will be instructed to wear it on the waist band above the hip during all waking hours and daily physical activity. The only exceptions would be when they are immersed in water (bathing or swimming) or in bed at night. They will also be instructed to reset the pedometer to zero at the beginning of each day and remove it at the end of the day. They will be given physical activity diary in which they will be asked to record: the time the pedometer was attached, removed and total number of steps displayed on the pedometer at the end of each day.During the fourth education session, i.e. one month after beginning the programme, participants will be asked to add strength exercises to their programme. The strength exercises will be performed at home and will be encouraged to keep a record in the physical activity diary: time, duration and any barriers to performing the exercise and how these were overcome. According to the United Kingdom physical activity guidelines and Start Active, Stay Active 2011, strength exercises for the major muscles of the lower limb, trunk and upper limb will be performed at home twice a week 8-12 repetitions of each exercise.

At the end of the study participants within the intervention group will keep the pedometer, as thanks for enrolling in this study.

Participants will attend six weekly sessions in small groups of up to six people; the content of the sessions will be based on educational cognitive behavioural programme development, which will allow participants to challenge their way of thinking, and change negative coping skills, cognition and emotions. Each session will last approximately one hour, will be interactive, and will take place in the hospital. During the one hour education session,topics will be discussed as interactive session, with the physiotherapist and participants. Visit 1 will be a measurement session, the education sessions will start at visit 2, and all participants in the intervention group will receive a pedometer and information regarding how the pedometer should be used and physical activity diary which they will start to use.

In addition, participants will receive education material in the first education session visit 2, which will consist of written information describing the importance of both walking and a healthy diet for health benefits and the reduction of cardiovascular risk and other co- morbidities of RA. Education sessions and the written material will be in large text and be suitable for any reading age.

The intervention group will receive two booster sessions, after 3 and 6 months to provide support to the participants First session interactive discussion on cardiovascular disease (CVD), Rheumatoid arthritis, Risk of CVD in Rheumatoid Arthritis, the importance of physical activity, Goal setting, instruction and practice on how to use pedometer.

second session Group discussion regarding exercise and physical activity and self-monitoring of behaviour, barriers to physical activity (Problem solving), advice, discussion on the importance of social support.

session 3 Relapse prevention, Control over CVD via lifestyle behaviour. session 4 Relevance and importance of strength training and opportunity to practice exercises.

session 5 Interactive discussion regarding healthy diet, strategies to enhance perceived control.

session 6 Motivation, Social facilitation, Action planning for the next 6 weeks.

First booster session Discuss any barriers, encouragement and motivation of the participants to continue in this programme.

Second Booster session Discuss any barriers, encouragement and motivation of the participants to continue in this programme.

Comparison Group The comparison group will be assessed at baseline (visit1), , after they have agreed to enroll in this study. The assessment will take approximately one hour; participants randomly allocated to the comparison group will receive one education session (visit 2) regarding the importance of exercise and healthy diet and will be given education material similar to intervention group and encouraged to read it. The comparison group will also be assessed at 3, 6 and 12 months (end of the study). On completion of the study all participants in the comparison group will be given a pedometer, activity diaries and advice on how to use them.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Rheumatoid Arthritis according to American College of Rheumatology (ACR)/ European League Against Rheumatism criteria (EULAR) 2010.
* Diagnosed within the first five years of disease.
* Willing and able to give written informed consent.
* Age 18 years and over.

Exclusion Criteria:

* Patients will be excluded, if they suffer from severe hypertension, joint replacement in the previous 6 months, unstable cardiac conditions and other serious pathology which would affect their ability to take part in physical activity such as uncontrolled diabetes.
* Pregnancy.
* Unable to understand written and spoken English.
* Cognitive impairment determined by the clinical judgment of the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity will be assessed.( ActivPAL monitor and International Physical Activity Questionnaire (IPAQ)) | Baseline, 3, 6 months and one year
  The measure is a composite. Objectively measured physical activity and sedentary behavior will be assessed using an ActivPAL activity monitor, which measures the posture and classifies daily living activity into periods spent sitting, lying, standing and stepping. An ActivPAL monitor will be used in assessment for 7 consecutive days to monitor individual physical activity, time spent sedentary and will also be used at each follow up assessment. The monitor will be attached to the participant's thigh at each assessment point and, following the seven day period.
  IPAQ is categorized into low, moderate and high physical activity.

SECONDARY OUTCOMES:
Change in RA assessment from baseline to end of the study using (Disease activity A simplified Disease Activity Index (SDAI) and Rheumatoid Arthritis Quality of Life (RAQoL)) | baseline, 3, 6 months and one year
  The measure is a composite.A simplified Disease Activity Index (SDAI) will be used to assess clinical disease activity based. The SDAI score is based on joint tenderness, swelling, patient global score (0-10), provider global score (0-10) and C - reactive protein mg/dl. The RAQoL is a self-assessment questionnaire score originally developed in the UK and the Netherlands. It consists 30 items with a yes/no (1/0) response format. The overall score is the sum of individual item scores the sore range from0-30 and the higher the score the poorer the quality of life.The questionnaires will be completed, face to face, during the assessments.
change in RA assessment from baseline to the end of the study Functional ability (Six minute walk test (6MWT),Stanford Health Assessment in functional capacity Questionnaire (HAQ) and Hand grip strength ) | baseline, 3, 6 months and one year
  The measure is a composite.The participants will be asked to walk for a period of six minutes, at their own pace, along a straight, 30 m hallway. Participants will be asked to cover as much ground as possible in six minutes, but will be allowed to stop if required. The distance in meters will be recorded at the end of the six minutes. A Health Assessment Questionnaire will be used to measure the capacity to perform activities in daily life. The score ranges from 0-3, with the higher score (3) indicating more disability and the lowest score (0) indicating no physical disability.The hand grip test will be done while the participant is in a sitting position with shoulders adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral and wrist between 0 and 30° of extension. The test will be repeated 3 times with the dominant hand, and maximum reading will be taken.
  The questionnaires will be completed, face to face, during the assessments.
change in Cardiovascular risk factors(Blood pressure will be measured,blood sample will be taken).Anthropometric variables Body mass index, waist circumference, waist hip ratio and waist height ratio. | baseline, 3, 6 months and one year
  The measure is a composite.Blood pressure will be measured. Routine clinical blood samples will also be taken in order to asses for lipids (e.g. total and HDL cholesterol and triglycerides), glucose, insulin, HbAlc, liver function (ALT, GGT, AST), inflammatory biomarkers (e.g. CRP), and NMR metabolomics profile (non- routine).
change in Dietary assessment(Dietary Instrument for Nutrition Education (DINE)) | baseline, 3, 6 months and one year
  The DINE method is a brief and inexpensive tool for diet assessment in primary care health promotion programmes.The DINE consists of questions regarding eating and drinking over the last 7 days, and scores are obtained for fatty and sugary food and fruit and vegetable intake.The questionnaires will be completed, face to face, during the assessments.
Change in Self-efficacy to Regulate Exercise | baseline, 3, 6 months and one year
  The Self-efficacy to Regulated Exercise questionnaire will be used, which is a reliable instrument with high internal consistency and satisfactory constructive validity (Kroll et al, 2007).The score ranges from 0-100 with the higher score (90-100) indicating high certainty and the lowest score (0) indicating cannot do.The questionnaires will be completed, face to face, during the assessments.
Change in Charlson Comorbidity Index | baseline, 3, 6 months and one year
  Charlson comorbidity index is a valid and reliable method of measuring comorbidity that can be used in clinical research. The score is reached by adding the comorbidity score to age score. The information will be taken from participant medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PhD, Study Director — University of Glasgow
Locations (1):
- Western Infimary, Glasgow, Glasgow, UK, United Kingdom